CLINICAL TRIAL: NCT02668094
Title: The Effect of Pregabalin on Pain of Propofol Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015-03-037-001
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Pain
Keywords: propofol; lidocaine; pregabalin
MeSH Terms: conditions — Pain | interventions — Lidocaine; Pregabalin; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group L (Active Comparator): Lidocaine 40mg was given intravenously before injection of propofol
  Interventions: Drug: Lidocaine; Drug: propofol
- Group LP (Active Comparator): Pregabalin 75 mg was given orally 2 hour before surgery
  Interventions: Drug: Pregabalin; Drug: propofol
- Group HP (Active Comparator): Pregabalin 150 mg was given orally 2 hour before surgery
  Interventions: Drug: Pregabalin; Drug: propofol

INTERVENTIONS:
Drug: Lidocaine
  Arms: Group L
Drug: Pregabalin
  Arms: Group HP; Group LP
Drug: propofol

SUMMARY:
Pain is a common side effect of propofol injection. The purpose of this study was to compare the efficacy of pregabalin and lidocaine in reducing propofol injection pain.

DETAILED DESCRIPTION:
In a randomized, double blind, prospective trial, 120 patients were allocated to one of three groups (each n=40) receiving intravenous lidocaine 40mg (group L), oral pregabalin 75 mg (group LP), and oral pregabalin 150 mg (group HP) as pretreatment, followed by injection of 25% of 2 mg/kg propofol. Pain was assessed by a four point scale (0=no, 1=mild, 2=moderate, 3=severe pain).

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent elective dental surgery.

Exclusion Criteria:

* Patient with a history of adverse response to lidocaine or pregabalin,
* Patient with cardiovascular or respiratory disease,
* Patient who takes any sedatives, analgesics, or anticonvulsants within 24 hours before surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Propofol injection pain | 10 seconds after injection of propofol
  Thirty seconds after pretreatment, 25% of the total calculated dose of propofol (2 mg/kg) was administrated into a dorsal hand vein. Ten seconds after injection of propofol, pain was assessed on a four-point scale (0=none, 1 = mild, 2= moderate, 3= severe).

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Dr, Principal Investigator — Kyungpook National Hosptial
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No